CLINICAL TRIAL: NCT02937285
Title: National Multicenter, Controlled, Single-blind Study With Two Parallel Groups Evaluating the Safety and Efficacy of Sequential Treatment With Mitoxantrone and Interferon Beta-1a (REBIF 44mg 3 Times / Week) Versus Interferon Alone in Patients With Strong Risk of Progression in the Initial Phase of Multiple Sclerosis
Brief Title: National Multicenter, Controlled, Single-blind Study With Two Parallel Groups Evaluating the Safety and Efficacy of Sequential Treatment With Mitoxantrone and Interferon Versus Interferon Alone in Patients With Strong Risk of Progression in the Initial Phase of Multiple Sclerosis
Acronym: MITOX-REBIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC10_8918; 2004-001601-10 (EudraCT Number)
Record Dates: First submitted 2016-09-09; First posted 2016-10-18 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a; Mitoxantrone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Interferon alone
  Interventions: Drug: Interferon beta 1a
- Experimental group (Experimental): Mitoxantrone for 6 month followed by interferon
  Interventions: Drug: Interferon beta 1a; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Interferon beta 1a — Subcutaneous injection of 44µg 3 times a week
  Other Names: REBIF
Drug: Mitoxantrone — 10 mg / m² monthly infusion for 6 months
  Other Names: ELSEP
  Arms: Experimental group

SUMMARY:
The relative effectiveness of current treatments and their different mechanisms of action yield to consider more and more that the multiple sclerosis (MS) therapeutic approach must use multiple molecules, both combined and sequential.

In this sense, one can assume that the combination of two molecules with different but complementary mechanisms of action, can delay progression of the disease. Mitoxantrone has a powerful action, immediate and total, whereas interferon a selective action, immunomodulatory and delayed.

DETAILED DESCRIPTION:
This study is based on the hypothesis that there is a synergistic effect of both increasing the dose of interferon and also the use of mitoxantrone, allowing to further reduce the conversion rate MS.

Because mitoxantrone decreases the rate of relapses 2 times more than interferon beta, a (at least) 2 times higher benefit on the disease activity is expected with interferon mitoxantrone combination than with interferon alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a MS according to the McDonald criteria:
* One relapse with time dissemination shown by an MRI performed less than 2 months before inclusion, with at least one of these criteria:
* multifocal presentation
* relapse determining a severe disability (EDSS greater than 3.5)
* at least 2 lesions taking contrast on MRI
* at least 9 T2 lesions with contrast enhancement.
* Patients must be 18 to 50 years.
* The duration of disease progression should be less than one year.
* Women of childbearing age must have an effective contraception.
* Patients have to be able to give their own informed consent before inclusion in the study.

Exclusion Criteria:

* presence of another disease that could explain the symptoms / signs of the patient.
* Any other condition / disability that may interfere with the clinical state.
* Prior treatment with immunosuppressive (mitoxantrone, azathioprine, cyclophosphamide) or immunomodulator.
* Treatment with corticosteroids in the previous 2 weeks, regardless of the dose.
* Corticosteroids for over a month.
* Pregnancy and lactation.
* Patient whose antecedents may contra-indicate the use of immunosuppressive therapy.
* Hypersensitivity to mitoxantrone or one of the excipients.
* Clinical cardiac disease with reduced ejection fraction of the left ventricle.
* Patient suffering from myelodysplasia.
* Abnormalities of Complete Blood Count.
* History of hematologic malignancy.
* Hepatic impairment.
* Vaccination against yellow fever.
* Vaccination with an attenuated vaccine assets.
* Treatment with phenytoin or fosphenytoin.
* Hypersensitivity to interferon beta-1a natural or recombinant or any of the excipients.
* Current severe depression and / or suicidal thoughts.
* Uncontrolled epilepsy.
* History of addiction.
* A history of hypersensitivity to gadolinium, history of severe renal impairment
* Inability to undergo MRI (claustrophobia, tics, involuntary movements, tremor, etc.).
* Participation in another trial in the preceding 6 months or during the study.
* Minors, protected adults and persons deprived of their liberty.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-12-06 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy | Four years after inclusion
  Efficacy is judged based on
  * the absence of relapse within the 2 first years; AND
  * a disease progression as determined by an increase in the Expanded Disability Status Scale (EDSS) not greater than 1 during the 4 years treatment.

SECONDARY OUTCOMES:
Time to first relapse | From date of randomization until the date of first documented progression, assessed up to 4 years
Frequency of relapses in 2 years | Within two years following randomization
Frequency of relapses in 4 years | Within four years following randomization
Changes in the level of disability in 2 years | Two years following randomization
  EDSS score
Changes in the level of disability in 4 years | Four years following randomization
  EDSS score
Patients in progression | Four years following randomization
  Rate of patients who progressed to a clinically definite MS (according to the criteria of Mc Donald) in the subgroup of patients who had only one clinical event.
Disease activity on MRI at 6 months | 6 months following randomization
  To compare in the two arms, the rate of patients without radiological (MRI) sign of disease activity
Patients without disease activity on MRI at 12 months | 12 months following randomization
  To compare in the two arms, the rate of patients without radiological (MRI) sign of disease activity
Patients without disease activity on MRI at 24 months | 24 months following randomization
  To compare in the two arms, the rate of patients without radiological (MRI) sign of disease activity
Patients without disease activity on MRI at 48 months | 48 months following randomization
  To compare in the two arms, the rate of patients without radiological (MRI) sign of disease activity
Number of visible lesions on MRI at 6 months | 6 months following randomization
  To compare in the two arms, the number of lesions taking contrast
Number of visible lesions on MRI at 12 months | 12 months following randomization
  To compare in the two arms, the number of lesions taking contrast
Number of visible lesions on MRI at 24 months | 24 months following randomization
  To compare in the two arms, the number of lesions taking contrast
Number of visible lesions on MRI at 48 months | 48 months following randomization
  To compare in the two arms, the number of lesions taking contrast
Lesion load on evaluated T2 weighted MRI at 12 months | 12 months following randomization
Lesion load on evaluated T2 weighted MRI at 24 months | 24 months following randomization
Lesion load on evaluated T2 weighted MRI at 48 months | 48 months following randomization
Brain atrophy | 24 and 48 months following randomization
  To assess the presence and progression of brain atrophy, changes in the total brain volume after 24 and 48 months will be automatically measured from MR images with dedicated software and expressed as percent change, from a standardized estimation of cerebral volume.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles EDAN, MD, PhD, Study Director — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No